CLINICAL TRIAL: NCT03389295
Title: Sequential Chemoradiotherapy With Reduced Target Delineation and Radiation Doses During Radiotherapy for Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Reduced Target Delineation and Radiation Doses Chemoradiotherapy for Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiayun He, MD (Other)
Responsible Party: Sponsor-Investigator, Xiayun He, MD, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPF-Shanghai
Record Dates: First submitted 2017-12-20; First posted 2018-01-03 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Reduced Target Delineation and Radiation Doses; Sequential chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: Drug: TPF regimen comprised docetaxel (60 mg/m2/day, day 1), cisplatin (25 mg/m2/day, days 1-3), and 5-fluorouracil (500 mg/m2/day with a 120-h infusion) Radiotherapy：Reduced Target Delineation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reduced Target Delineation and Radiation Doses (Experimental): All patients were assigned to receive induction chemotherapy (IC) followed by IMRT with adjuvant chemotherapy (AC). IMRT was administered 2 weeks after IC, and AC was administered 1 month after IMRT. IC or AC (TPF regimen) comprised docetaxel (60 mg/m2/day, day 1), cisplatin (25 mg/m2/day, days 1-3), and 5-fluorouracil (500 mg/m2/day with a 120-h infusion) administered once every 3 weeks for two cycles. During radiotherapy, involved retropharyngeal lymph nodes and intracavity lesions of the primary tumor were delineated according to the post-IC volume, whereas the remainder of the involved tissues (eg, pterygopalatine fossa) of the primary tumor were delineated according to the pre-IC volume of the primary tumor as shown by MRI. Post-IC volumes of involved neck lymph nodes were used for delineation. The prescribed dose was 66 Gy to tumors above the slices of skull base or below the orapharynx with less than 5 mm retropharyngeal lymph nodes, or 70.4 Gy to tumors in other slices.
  Interventions: Radiation: Reduced Target Delineation and Radiation Doses

INTERVENTIONS:
Radiation: Reduced Target Delineation and Radiation Doses — The target volumes were delineated according to the treatment protocol defined as follows: the GTV of the primary tumor (GTV-P) included retropharyngeal lymph nodes, considering the common phenomena of integration, and the rest involved lymph nodes that were defined as GTV-N. For the GTV-P, involved retropharyngeal lymph nodes and intracavity lesions were delineated according to the post-IC volume, whereas the remainder of the involved tissues (eg, pterygopalatine fossa) were delineated according to the pre-IC volume of the primary lesion as shown by MRI. Post-IC volumes of involved neck lymph nodes were used for GTV-N delineation.
  The prescribed dose was 66 Gy to tumors above the slices of skull base or below the orapharynx with less than 5 mm retropharyngeal lymph nodes, or 70.4 Gy to tumors in other slices.
  Other Names: Drug: TPF regimen comprised docetaxel (60 mg/m2/day, day 1), cisplatin (25 mg/m2/day, days 1-3), and 5-fluorouracil (500 mg/m2/day with a 120-h infusion)

SUMMARY:
To determine the efficacy and safety of sequential chemoradiotherapy with regimen of docetaxel, cisplatin and fluorouracil and reduced target delineation and radiation doses IMRT for patients with locoregionally advanced nasopharyngeal carcinoma

DETAILED DESCRIPTION:
Although concurrent chemoradiation is the standard treatment modality for locally advanced nasopharyngeal carcinoma (NPC), high incidences of distant metastases and severe treatment related toxicities have become an obstacle to be overcome. Besides, a common problem in locally advanced NPC is the narrow gap between the tumor and critical normal structures, which makes dose optimization difficult. Considering that significant tumor shrinkage may occur during induction chemotherapy, and incidences of distant metastases may be reduced by adjuvant chemotherapy, this study was designed to explore the efficacy and safety of sequential chemoradiotherapy with regimen of docetaxel, cisplatin and fluorouracil and reduced target delineation and radiation doses IMRT for patients with locoregionally advanced NPC.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically proven nasopharyngeal carcinoma (WHO type 2 or 3)
2. Stage Ⅲ-ⅣB disease (AJCC/UICC 2010)
3. KPS more than 70
4. Life expectancy of more than 6 months
5. Signed written informed consent
6. Adequate organ function including the following:

Absolute neutrophil count (ANC) >= 1.5 * 109/l Platelets count >= 100 * 109/l Hemoglobin >= 10 g/dl AST and ALT <= 2.5 times institutional upper limit of normal (ULN) Total bilirubin <= 1.5 times institutional ULN Creatinine clearance >= 50 ml/min Serum creatine <= 1 times ULN

Exclusion Criteria:

1. Evidence of distant metastasis
2. Prior chemotherapy or anti-cancer biologic therapy for any type of cancer, or prior radiotherapy to the head and neck region
3. Other previous or concomitant cancer, except for in situ cervical cancer and cutaneous basal cell carcinoma
4. Pregnant or breast-feeding females, or females and males of childbearing potential not taking adequate contraceptive measures
5. Presence of an uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | up to 5 years
  The time from date of treatment until date of first documented disease progression or death from any cause, assessed up to 5 years.

SECONDARY OUTCOMES:
Local recurrence-free survival | up to 5 years
  The time from date of treatment until date of first documented disease recurrence at a local site, assessed up to 5 years.
Regional recurrence-free survival | up to 5 years
  The time from date of treatment until date of first documented disease recurrence at a regional site, assessed up to 5 years.
Overall survival | up to 5 years
  The time from date of treatment until date of death due to any cause, assessed up to 5 years.
Distant metastasis-free survival | up to 5 years
  The time from date of treatment until date of first documented distant metastasis, assessed up to 5 years.
Locoregional failure patterns | up to 5 years
  The failures were categorized as occurring inside or outside the high dose target volume, depending on the location of Vrecur: "in field" if 95% of Vrecur was within the 95% isodose; "marginal" if 20% to 95% of Vrecur was within the 95% isodose, or "outside" if less than 20% of Vrecur was inside the 95% isodose.
Number of participants with acute toxicities | during treatment
  Number of participants with acute toxicities occurred during the chemoradiotherapy according to CTCAE4.0
Number of participants with late toxicities | up to 5 years
  Number of participants with late toxicities occurred from 3 months after completion of radiotherapy to last follow-up visit according to Radiation Therapy Oncology Group radiation morbidity scoring criteria.
Changes of tumor volume | 2 weeks after completion of induction chemotherapy
  Changes of tumor volume before and after induction chemotherapy
Relationship between treatment failure and dose received by target | up to 5 years
  Relationship between treatment failure and dose received by target

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xue F, Ou D, Ou X, Zhou X, Hu C, He X. Long-term results of the phase II dose and volume de-escalation trial for locoregionally advanced nasopharyngeal carcinoma. Oral Oncol. 2022 Nov;134:106139. doi: 10.1016/j.oraloncology.2022.106139. Epub 2022 Sep 27. PMID 36179488